CLINICAL TRIAL: NCT05450614
Title: Smartphone App Based Cognitive Behavioral Therapy Versus Online Group Cognitive Behavioral Therapy: Randomized, Non-inferiority Clinical Trial
Brief Title: Smartphone App Based CBT Versus Online Group CBT: Randomized, Non-inferiority Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200484
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major; Cognitive Behavioral Therapy; Clinical Trial; Smartphone; Machine Learning
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Initially, patients who accept the invitation will be randomized between groups Thrive vs CBCT. In the Thrive group, access to the application and information regarding its use will be made available to participants. Reassessments and data collection will be performed at 5 points: baseline, 4, 8, 12 weeks and 6 months. These five evaluations will be carried out through questionnaires sent to the participants. Participants selected for the TCCG group will undergo a new randomization, which will select 50% of patients for immediate start of online sessions and the remainder for inclusion in a waiting list. Participants selected for immediate start will start the CBCT sessions at the time of the initial assessment and will be reassessed at the same points as the Thrive group, also through self-administered online questionnaires. A 12-week assessment list through online auto scales will take place at the end of the period. Patients at PHQ≥ 9 will initiate CBCT protocol sessions online.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrive app (Experimental): In the Thrive group, access to the application and information regarding its use will be made available to participants. Reassessments and data collection will be performed at 5 points including baseline, 4 weeks, 8 weeks, 12 weeks and 6 months. These five evaluations will be carried out through questionnaires sent to the participants.
  Interventions: Other: Thrive app
- TCCG (Active Comparator): Participants selected for the TCCG group will undergo a new randomization, which will select 50% of patients for immediate start of online sessions and the remainder for inclusion in a waiting list. Participants selected for immediate start will start the CBCT sessions at the time of the initial assessment and will be reassessed at the same points as the Thrive group, also through self-administered online questionnaires.
  The waiting list will last for 12 weeks, with assessment through self-applicable online scales at the end of the period. Patients who present PHQ≥ 9 will then start online CBCT sessions, according to the protocol above.
  Interventions: Behavioral: TCCG

INTERVENTIONS:
Other: Thrive app — The application has already been developed using the Flutter framework and provides users with the main CBT-based strategies to reduce depressive symptoms. In order to engage users, gamification strategies were also implemented. Some examples are 1) development and achievement: quiz on psychoeducation with rewards; 2) epic sense: like the messages in the psychoeducation session; 3) unpredictability: surprise quiz. An avatar will also be available for the participant, who will gain experience as he interacts with some of the application's functions. Finally, participants will receive weekly videos of less than 5 minutes with tips on how to use the app. There will be a total of 12 videos with psychoeducation tips and how to use the application.
  Arms: Thrive app
Behavioral: TCCG — In the literature, there is no single protocol for the treatment of depression through CBCT, therefore, a systematized protocol was developed for this study, aiming to structure and unify this intervention. Participants selected for the TCCG group will be randomly divided into 10 groups of 10 members each. The TCCG will be held through weekly meetings, exclusively online. Twelve sessions lasting 90 minutes each will be applied. The structuring of the sessions is based on the cognitive-behavioral model, starting with psychoeducation about the disorder and self-knowledge, starting with cognitive restructuring and relapse prevention. Homework will be part of the protocol. The sessions will be held on a digital platform (Google Meet) and access instructions will be provided to the participants of this group in the evaluation interview.
  Arms: TCCG

SUMMARY:
The present research project aims to compare the efficacy and safety of an intervention based on a smartphone application, which uses CBT techniques, to online group cognitive behavioral therapy (CBCT), in improving depressive symptoms.

The project also has supplemental analysis to predict who will respond to the CBT intervention using the application. For this analysis, machine learning algorithms, a set of techniques from the field of artificial intelligence, will be used to create a predictive calculator for response to interventions. The analysis protocol used for this analysis will be in accordance with that proposed in task Force of the International Society for Bipolar Disorders.

DETAILED DESCRIPTION:
This is a randomized, non-inferiority, three-arm clinical trial, one of which consists of a waiting list. Participants in this study will be selected from an online survey already carried out and approved by the National Research Ethics Committee (Conep), which included 5,000 participants. Patients will be randomized to one of the study arms, application (Thrive) or CBCT (immediate start versus waiting list). Digital interventions in mental health have been gaining strength in the scientific literature, and recently the US Food and Drug Administration (FDA) authorized the digital prescription of an app to treat insomnia. This type of intervention is not a substitute for clinical consultation, but it can be useful in circumstances related to poor access to mental health services, which is a chronic problem in many developing and underdeveloped countries, but which has been exacerbated recently with the COVID-19 pandemic. 19. Of note, CBT is a first-line treatment for combating depressive symptoms, and its use has recently been studied on digital platforms. To help participants in this stage and increase their engagement, the app will provide access to a virtual caregiver and gamification strategies as reported in a recent editorial published in a famous scientific journal.

For this clinical trial, 400 participants with the expected symptoms among those who responded to the aforementioned clinical trial will be invited to be surveyed (National Trial Committee Survey Approved in Research Conducted and Approved).

The goals of this article will not be carried out in the main scientific journals of medicine, but also to assess whether a low-cost digital intervention designed only for reviews where the improvement in mental health is low may the altered symptoms of the included access . It is important that this intervention is useful not only in periods of social isolation, but also when the pandemic ends, since 1) about 50% of patients with depression do not have consultations with mental health professionals; 2) we expect an increase in the number of people with depression after the pandemic, due to its consequences.

Our hypothesis is that the smartphone application, with CBT techniques, although it does not replace the face-to-face consultation, is safe and is not inferior to the CBCT. If shown to be effective, this app will be an innovative, low-cost strategy for dealing with depressive symptoms during and after the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* have depressive symptoms characterized by PHQ-9≥9 and a diagnosis of Major Depressive Episode through the Mini-International Neuropsychiatric Interview instrument -- own a smartphone
* agree with the treatment objectives and sign the consent form
* age between 18 and 65 years
* be living in Brazil and be fluent in Portuguese.

Exclusion Criteria:

* pregnancy
* initiation of any psychological treatment within the previous 3 months
* visual impairment that prevents use of the app
* current risk of suicide
* bipolar disorder, schizophrenia, schizoaffective disorder, intellectual disability, and alcohol or drug abuse in the last year.

Other comorbid medical conditions will also be included, unless they are degenerative (dementia or multiple sclerosis) in a way that could compromise interaction with the application. Participants may be taking psychotropic drugs, including medication for depression, if the medication regimen has not changed in the previous 3 months and if there has been no change over the course of study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
reduction of Patient Health Questionnaire (PHQ-9) averages | week 12
  reduction of PHQ-9 averages. PHQ >= 9 indicates positive screening for current depressive episode.

SECONDARY OUTCOMES:
reduction of anxiety symptoms | week 12
  measured by the Generalized Anxiety Disorder Screener (GAD-7). It consists of seven items, arranged on a four-point scale: 0 (never) to 3 (almost every day), with a score ranging from 0 to 21, when measuring the frequency of signs and symptoms of anxiety in the last two weeks. . A positive indicator of signs and symptoms of anxiety disorders is considered to be a value equal to or greater than 10.
adherence of the participants to the app | access for at least 15 minutes per week
  In the Thrive app group, accessing, for at least 15 minutes per week, the app will be considered a membership criterion; in the TCCG group, participation in the sessions will be the adhesion criterion, with a maximum of 4 absences being tolerated.
levels of loneliness | week 12
  measured by the UCLA loneliness scale (UCLA) - brief version of 3 items

CONTACTS AND LOCATIONS:
Overall Officials: Ives C Passos, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil

REFERENCES:
- [Derived] Bebber JC, Braga Montezano B, de Souza Vivan A, Antonelli-Salgado T, Aguiar KR, Zimerman A, Shintani AO, Braga Ryff Moreira M, Campos R, Rodrigues L, Frisina Zaffari G, Mallmann G, Fernandes Pulice R, Chiodelli Senger V, Rosendo Vargas J, Zimmer C, Dos Santos Amaral MC, Goncalves Veloso G, Dalla Vecchia GF, Bisognin Lopez JC, Brunoni AR, Rabelo-da-Ponte FD, Passos IC, Braga DT. Digital interventions for depressive symptoms: a randomized clinical trial. Trends Psychiatry Psychother. 2025;47:e20241006. doi: 10.47626/2237-6089-2024-1006. Epub 2025 May 11. PMID 40349367